CLINICAL TRIAL: NCT06135337
Title: A Prospective, Exploratory, Randomized, Subject- and Evaluator - Blinded, Parallel- Group, Single-centre, Pilot Trial Investigating the Safety and Effect of THIODERM ELATE Compared to Juvéderm® Ultra 3 for Lip Augmentation (TILI)
Brief Title: THIODERM ELATE for Augmentation of Very Thin, Thin, and Moderately Thick Lips
Acronym: TILI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Croma-Pharma GmbH (Industry)
Collaborators: Proinnovera GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPH-70601
Record Dates: First submitted 2023-11-10; First posted 2023-11-18 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Lip Abnormality
Keywords: Lips; Volume Deficit; Hyaluronic Acid; Dermal Filler

STUDY DESIGN:
Intervention Model Description: Parallel-Group Design with random assignment to test device or comparator device in a 2:1 ratio
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects and Evaluating Investigator will be blinded to study device assignment. The subject will be blind-folded during treatment. The Evaluating Investigator is unaware of the device assignment and has no access to study data that could potentially contain unblinding information
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group THIODERM ELATE (Experimental): Subjects who will receive THIODERM ELATE into upper and lower lip (66.7% of enrolled subjects)
  Interventions: Device: Thioderm Elate
- Group JUVÉDERM ULTRA 3 (Active Comparator): Subjects who will receive JUVÉDERM ULTRA 3 into upper and lower lip (33.3% of enrolled subjects)
  Interventions: Device: Juvéderm Ultra 3

INTERVENTIONS:
Device: Thioderm Elate — Test Device
  Arms: Group THIODERM ELATE
Device: Juvéderm Ultra 3 — Active Comparator Device
  Arms: Group JUVÉDERM ULTRA 3

SUMMARY:
This mono-center clinical investigation is intended to assess the safety and effectiveness of THIODERM ELATE for augmentation of very thin and thin lips in comparison with Juvéderm® Ultra 3.

DETAILED DESCRIPTION:
The Investigation is a prospective, exploratory, randomized, subject and evaluator - blinded, parallel-group, single-centre, pilot trial investigating the safety and effectiveness of THIODERM ELATE compared to Juvéderm® Ultra 3 for lip augmentation. Up to 33 eligible subjects will be included in this investigation with a 10 % estimated drop-out rate and will be randomized in a 2:1 ratio to Thioderm ELATE and Juvéderm® Ultra 3, respectively, after the informed consent form (ICF) has been signed and relevant pre-treatment procedures, including medical history and pregnancy testing, as well as eligibility for inclusion have been performed. Subjects will receive injections into both, upper and lower lip using Thioderm ELATE or Juvéderm® Ultra 3 until an optimal cosmetic result is achieved. During Screening and prior to injection, the Blinded Evaluating Investigator will evaluate the lip fullness by using the 5-point Lip Fullness Scale (LFS). An optional touch-up treatment can be performed at Week 4 upon discretion of the treating investigator. The safety and effectiveness of the treatment will be evaluated after Day 1, 3 and 7 as well as at 4, 8,12, 16 and 24 weeks or an End of Study Visit using objective and subjective outcome parameters. . The same Blinded Evaluating Investigator will assess each subject at screening and at the follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years at the time of screening (upper limit 75 years, inclusive).
2. Subjects with approximately symmetrical 'very thin' or 'thin' lips (scores of 1 or 2 on the 5-point Lip Fullness Scale) as assessed by the Blinded Evaluating Investigator at Screening (Visit 0). The scores do not have to be the same on both (upper and lower) lips, but must be 1 or 2.
3. Healthy skin in the perioral area and free of diseases that could interfere in cutaneous aging evaluation.
4. Intact or permanently replaced central and lateral incisors, canine and first and second premolars in the upper row of teeth and intact or replaced incisors, canines and premolars in the lower row of teeth
5. Subject has a stable medical condition with no uncontrolled systemic disease.
6. Females of childbearing potential must have a negative urine pregnancy test and must agree to use a highly effective method of birth control throughout the entire study.
7. Male subjects with female partners of child-bearing potential must agree to use contraception throughout the entire study (surgical sterilization or a physical barrier such as a condom).
8. Willingness to abstain from any aesthetic or surgical procedures in the treatment area for the duration of study, including botulinum toxin injection (except glabella or forehead botulinum toxin treatment).
9. Subjects who understand the purpose and conduct of the study and having given written informed consent and are willing and able to attend the study visits as judged by the Investigator.

Exclusion Criteria:

1. Females, who are pregnant and/or, lactating or planning to become pregnant during the clinical investigation.
2. History of allergies or hypersensitivity to hyaluronic acid and/or to gram positive bacterial proteins, lidocaine or any amide-based anaesthetic
3. History of severe allergies manifested by a history of anaphylaxis or history or presence of multiple severe allergies
4. Tendency to keloid formation and/or hypertrophic scars.
5. Presence of infectious, inflammatory or proliferative cancerous or pre-cancerous lesions in the area to be treated
6. Recurrent (three times a year over the last year) herpes simplex in the treatment areas
7. Known human immune deficiency virus-positive individuals
8. History or presence of any autoimmune or connective tissue disease
9. Uncontrolled (or unstable) Diabetes mellitus or uncontrolled systemic diseases as per Investigator discretion
10. Previous facial plastic surgery, tissue augmentation with silicone, fat or another non-absorbable substance (permanent fillers) and semi-permanent / long-lasting fillers (e.g., poly-L-lactic acid (PLLA), Polymethylmethacrylate (PMMA) filler) in the area of device application and during the entire investigation
11. Implantation of dermal fillers in the treatment area within the preceding 24 months prior to Visit 0 (Screening) and during the entire investigation
12. Subject has received any of the following aesthetic treatments in the perioral area and or lower face third: e.g., laser therapy, absorbable and non-absorbable sutures (threads), dermabrasion, mesotherapy, micro-needling and/or botulinum toxin (including treatment of crow´s feet in the outer eye region) as well as permanent make-up at the lips within the last 12 months prior to Visit 0, chemical peeling within the last three months prior to Visit 0 or is planning to undergo such procedures during entire investigation
13. Facial lipolysis, including submental fat treatments, within the previous 12 months prior to Visit 0 (Screening) and during the entire investigation
14. Bariatric surgery within 12 months prior to Visit 0 (Screening) and during the entire investigation.
15. History of bleeding disorder and/or use of anticoagulant, antiplatelet or thrombolytic medication from 10 days pre- to 3 days post-injection (initial treatment and touch-up treatment).
16. Systemic glucocorticoids, including immunosuppressant or immunomodulators, within 8 weeks prior to undergoing investigational device injections.
17. Subjects suffering from untreated epilepsy.
18. Subjects with acute rheumatic fever with heart complications.
19. Subjects with symptoms of cardiac conduction disorders.
20. Planned dental/oral surgery or modification (bridgework, implants) within four weeks prior to each injection and to a minimum of four weeks post injection (initial treatment, touch-up treatment).
21. Beard longer than three-day beard, or excessive facial hair that could interfere in evaluation of treatment as judged by the Investigator.
22. Subjects with active SARS-CoV-19 infection and Subjects with symptoms consistent with COVID-19 infection including any other respiratory symptoms/illnesses within the past 14 days unless tested negative prior to Visit 0 (Screening).
23. Any medical condition prohibiting the inclusion in the clinical investigation according to the judgment of the Investigator.
24. Previous enrolment in this clinical investigation.
25. Current participation in another clinical investigation, or treatment with any investigational drug/medical device within 30 days prior to clinical investigation enrolment, or 5 half-lives of the investigational drug, whichever is longer.
26. Subjects who experienced fat loss for a minimum of 10% of body weight over the last 12 months (e.g., post bariatric subjects), or Subjects who have the intention to change eating habits that result in a weight gain or loss >10% during the entire investigation.
27. Close affiliation with the Investigator (e.g., a close relative, financially dependent on the study site) or Subject who is an employee of the Sponsor's company or group companies of the Sponsor.
28. Any individual whose willingness to volunteer in this clinical investigation could be unduly influenced by the expectation, whether justified or not, of benefits associated with participation or of retaliatory response from senior members of a hierarchy in case of refusal to participate (e.g., persons with a legal custodian appointed due to mental disability, prisoners, soldiers and other members of the armed forces, civil servants).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Primary Safety Evaluation | through study completion, an average of 24 weeks
  Treatment-emergent AEs related to study treatment.

SECONDARY OUTCOMES:
Safety Evaluation | through study completion, an average of 24 weeks
  Frequency, severity, and causal relationship of adverse events (AEs) and serious adverse events (SAEs) during the entire study period, including adverse device effects (ADEs) and serious adverse device effects (SADEs)
Injection Site Reactions (ISR) | Week 1-4 (Week 1-8 in case of touch-up treatment)
  Injection site reactions as recorded in the Subject diaries during the first 4 weeks (28 days) after baseline- or touch-up-treatment. Injection site reactions will be assessed overall
Responder Rate Week 12 | Week 12
  Response measured on the 5-point LFS at Week 12 compared to baseline, based on the Blinded Evaluating Investigator's live assessment where responder is defined as a subject with a ≥1 improvement of the upper lip AND a ≥1 improvement of the lower lip
Required total Volume of Injection | Day 0; Week 4 (in case of touch-up treatment)
  Required total volume for optimum aesthetic result for treatment of the lip volume deficit at baseline and optional touch - up treatment at Week 4 of the upper and lower lip, as well as for the lip overall.
Responder Rate | Day7; Week 4, 8, 16, and 24 and at end of study
  Response measured on the 5-point LFS at Day 7 and Week 4, 8, 16, 24 and End of Study compared to baseline, based on the Blinded Evaluating Investigator's live assessment where a responder is defined as a Subject with a ≥1 improvement on the upper lip AND a ≥ 1 improvement on the lower lip on the 5-point LFS
Magnitude of Response Upper Lip (Investigator) | Day7; Week 4, 8, 12, 16, and 24
  Change of 5-point LFS of the upper lip from baseline to Day 7 and Week 4, 8, 12, 16, 24 and at End of Study based on the Blinded Evaluating Investigator's live assessment
Magnitude of Response Lower Lip (Investigator) | Day7; Week 4, 8, 12, 16, 24 and End of Study
  Change of 5-point LFS of the lower lip from baseline to Day 7 and Week 4, 8, 12, 16 and 24and at end of study based on the Blinded Evaluating Investigator's live assessment
Magnitude of Response Both Lips (Investigator) | Day7; Week 4, 8, 12, 16, 24 and End of Study
  Change of 5-point LFS of the overall lip from baseline to Day 7 and Week 4, 8, 12, 16 and 24 and at end of study based on the Blinded Evaluating Investigator's live assessment
Magnitude of Response Upper Lip (Independent Photo Review Panel) | Day7; Week 4, 8, 12, 16, and 24
  Change of 5-point LFS of the upper lip from baseline to Day 7 and Week 4, 8, 12, 16 and 24 based on the independent blinded evaluating panel's assessment
Magnitude of Response Lower Lip (Independent Photo Review Panel) | Day7; Week 4, 8, 12, 16, and 24
  Change of 5-point LFS of the lower lip from baseline to Day 7 and Week 4, 8, 12, 16 and 24 based on the independent blinded evaluating panel's assessment
Magnitude of Response Both Lips (Independent Photo Review Panel) | Day7; Week 4, 8, 12, 16, and 24
  Change of 5-point LFS of the overall lip from baseline to Day 7 and Week 4, 8, 12, 16 and 24 based on the independent blinded evaluating panel's assessment
Aesthetic Improvement (Investigator) | Week 4, 8, 12, 16, 24 and end of stidy
  Aesthetic improvement based on the Blinded Evaluating Investigator's assessment at Week 4, 8,12, 16 and 24 and at end of study using the GAIS
Aesthetic Improvement (Subject) | Week 4, 8, 12, 16, 24 and end od study
  Aesthetic improvement based on the Subject's assessment at Week 4, 8,12, 16 and 24 and at end of study using the GAIS
Lip Volume Change | Week 4, 8, 12, 16, 24 and end of study
  Volume change of the lips at Day 7 and Week 4, 8,12, 16 and 24 and at end of study, based on 3D surface imaging in comparison to the baseline 3D image
Subject's satisfaction (Outcome) | Day 1, 3, 7 and Week 4, 8,12, 16, 24 and end of study
  The extent of subject´s satisfaction with treatment of the lips at Day 1, 3, 7 and Week 4, 8,12, 16 and 24 and at ebd of study as assessed by the FACE-Q(TM) Satisfaction with Outcome Scale
Subject's satisfaction (Lips) | Day 1, 3, 7 and Week 4, 8,12, 16 24 and end of study
  The extent of subject´s appearance appraisal at Day 1, 3, 7 and Week 4, 8,12, 16 and 24 and at end of study as assessed by the FACE-QTM Satisfaction with Lip Scale
Pain Assessment | Day 0; Week 4 (in case of touch-up treatment)
  Subject´s pain assessment after each treatment on an 11-point scale, where 0 is no pain and 10 is the worst pain imaginable

CONTACTS AND LOCATIONS:
Locations (1):
- H&P Ambulatorien GmbH, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No